CLINICAL TRIAL: NCT06539598
Title: Impact of Respiratory Training in Swallowing and Respiratory Function in Patients With Friedreich's Ataxia
Brief Title: Respiratory Training in Friedreich's Ataxia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: IRB202401099
Record Dates: First submitted 2024-07-30; First posted 2024-08-06 (Actual); Last update posted 2025-11-03 (Actual); Status verified 2024-09

CONDITIONS: Friedreich Ataxia
MeSH Terms: conditions — Friedreich Ataxia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Respiratory Strength Training (RST) (Experimental): Participants will receive a respiratory strength training device to take home and use up to 5 times a week for 12 weeks.
  Interventions: Other: Respiratory Strength Training (RST)

INTERVENTIONS:
Other: Respiratory Strength Training (RST) — Respiratory Strength training involves inhaling/exhaling against a fix resistant to potentially increase respiratory strength

SUMMARY:
This is a prospective interventional study of patients with Friedreich's Ataxia that receive respiratory strength training for a period of 12 weeks with two research visits at the beginning and at the end of the study period. Visits include swallowing evaluation with fiberoptic endoscopic evaluation of swallowing, pulmonary function testing, surface electromyography and patient surveys.

ELIGIBILITY:
Inclusion Criteria:

* confirmed genetic testing of Friedreich's Ataxia
* have an overall DIGEST score of 1 or higher based on FEES screening
* are able to perform pulmonary function testing

Exclusion Criteria:

* have been on antibiotics within 15 days prior to baseline screening.
* have been prescribed systemic corticosteroids or neuromuscular blocking agents within 15 days of the baseline screening
* have an allergy or contraindication to topical lidocaine or oxymetazoline
* have any other concurrent medical condition which, in the opinion of the investigators, would make the subject inappropriate to participate in testing or respiratory exercise

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2024-08-29 (Actual); Primary Completion 2025-08-07 (Actual); Study Completion 2025-08-07 (Actual)

PRIMARY OUTCOMES:
Force Vital Capacity | Through study completion (4 months)
  Forced Vital Capicity will be measured before and after the 12 week intervention
Maximal Inspiratory Pressure (MIP) | Through study completion (4 months)
  Maximal Inspiratory Pressure (MIP) will be measured before and after the 12 week intervention
Maximal Expiratory Pressure (MEP) | Through study completion (4 months)
  Maximal Expiratory Pressure (MEP) will be measured before and after the 12 week intervention
Sniff Nasal Inspiratory Pressure (SNIP) | Through study completion (4 months)
  Sniff Nasal Inspiratory Pressure (SNIP) will be measured before and after the 12 week intervention
Swallowing | Through study completion (4 months)
  Fiberoptic Endoscopic Evaluation of Swallowing (FEES) will be measured before and after the 12 week intervention.
Surface Electromyography (sEMG) | Through study completion (4 months)
  sEMG will be placed on the skin to measure muscle activity involved in breathing and swallowing
Diaphragm Ultrasound | Through study completion (4 months)
  Diaphragm movement will be measured through an ultrasound probe positioned on the skin before and after the 12 week intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Carmen Leon Astudillo, MD, Principal Investigator — University of Florida
Locations (1):
- Clinical Research Center, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: No